CLINICAL TRIAL: NCT05152979
Title: Effects of On-line and In-clinic Intervention With Verb Network Strengthening Treatment (VNeST) on Word Finding in Aphasia
Brief Title: Effects of Verb Network Strengthening Treatment (VNeST) on Word Finding in Aphasia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After a pre study including two participants in a Single Case Research Design it was concluded that that the study design, needed to be slightly revised. A new registration has been submitted to the Clinical Trials, describing the new study design.
Sponsor: Göteborg University (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-02465
Record Dates: First submitted 2021-10-18; First posted 2021-12-10 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Anomia; Aphasia; Stroke
MeSH Terms: conditions — Anomia; Aphasia; Stroke

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Outcomes Assessor
Masking Description: The results are assessed by independent assessors blinded to in which phase (pre-post-follow up) the data is obtained, and partly to conditions for therapy (In-Clinic or Telepractice).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telepractice treatment (TP-T) (Experimental): Participants will receive 30 hours of training, 2-3 times a week in ten weeks using Verb Network Strengthening Treatment (VNeST).
  Treatment will be done with a speech-language pathologist providing the therapy through an online platform.
  Interventions: Behavioral: Verb Network Strengthening Treatment (VNeST)
- In-clinic treatment (IC-T) (Active Comparator): Participants will receive 30 hours of training, 2-3 times a week in ten weeks using Verb Network Strengthening Treatment (VNeST).
  Treatment will be done with a speech-language pathologist providing the therapy in person at a clinic.
  Interventions: Behavioral: Verb Network Strengthening Treatment (VNeST)

INTERVENTIONS:
Behavioral: Verb Network Strengthening Treatment (VNeST) — Participants are presented with a verb (representing an activity, for example, driving) orally and in writing. The participants are first asked to name someone who may perform the given activity (an agent, for example, a chauffeur), then to name an object which the given activity may be performed with (a patient, for example, a limousine). Several types of semantic clues and assistance are provided if the participant is having difficulties finding adequate nouns. This procedure is repeated for three different agents and objects related to the given verb. The participants are then asked to choose one of the three phrases participants have created and expand on it by telling where, when and why the agent is performing the activity. After this the participant are given sentences (with several foils) including the activity as well as agents and patients, and are asked to indicate whether the sentences are correct or not.

SUMMARY:
Although there is evidence that speech-language therapy may improve speech in language disorders following left hemisphere stroke there is still a lack of evidence for which types of therapy are effective. Furthermore, in Sweden, as well as in several other countries, access to speech-language therapy is limited. The purpose of this clinical trial is to compare outcome from Verb Network Strengthening Treatment (VNeST) provided as In-Clinic therapy (I-CT) or as synchronous telepractice therapy (TP-T).

DETAILED DESCRIPTION:
Every year thousands of persons in Sweden suffer from brain damage resulting in anomia, that is, word finding difficulties affecting their ability to talk to other people. Anomia is one of the most common and persistent symptoms of aphasia following a left hemisphere stroke, but it is also common in in progressive neurological diseases such as Parkinson's disease or multiple sclerosis (MS). There is evidence that more intensive speech language therapy may improve speech even in a chronic (> six month post stroke) phase of aphasia. However, access to the necessary amount of speech language therapy is limited due to lack of financial resources as well as to limitations to service providers in more rural areas.

It has been suggested that telepractice may increase the access to speech-language therapy for more people but there is a lack of knowledge of whether there is a difference in outcome from interventions provided as In-Clinic therapy (I-CT) or as telepractice therapy (TP-T).

Verb Network Strengthening Treatment (VNeST) is an anomia therapy focused on the production of short phrases. The participants generate thematically related verbs and nouns to strengthen the neural connections between the action (verb) and related thematic roles (agents and patients). From orally and written stimuli, the participants are asked to tell whom (subject) may do something (verb) with what (object) and then to do short expansions from this basic phrase. So far, results from single-case experimental design studies performed by Edmonds and colleagues are promising, showing generalization of outcomes to untrained items. Moreover, improvement in word finding was observed in other tasks like object and verb naming as well as sentence production and partly to connected speech.

The present project explores the effectiveness of VNeST, first in a small pilot study, then in a clinical trial including 80 participants. Participants with left hemisphere aphasia will be randomized to either an in-clinic therapy (I-CT) group or a telepractice therapy (TP-T) group and provided VNeST following the same treatment protocol based on Edmonds (2014).

Outcome measure include measures of naming ability on word- and phrase levels as well as in discourse. Measures of participant reported perceptions of functional communication and communicative participation as well as health related quality of life (PROMs) are also included.

ELIGIBILITY:
Inclusion Criteria:

* Aphasia and subjective experience of word finding difficulties
* Diagnosed left-hemisphere stroke at least six months post-onset
* With correction, sufficient hearing and vision to be able to participate in training and assessment
* Primarily speaking Swedish for at least the last 15 years

Exclusion Criteria:

* Other neurological injury or disease
* Moderately or severely impaired comprehension
* Moderate-severe apraxia of speech or dysarthria which may interfere with assessment
* Participation in any other speech-language treatment during the study
* Active substance dependence

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-01-16 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in naming ability of trained items at week 10. | Baseline, 10 weeks.
  Naming of ten trained phrases including an agent (subject), verb and a patient (object) with moving picture stimuli. Possible score ranges from 0 (worst) to 40 (best).
Change from baseline in naming ability of trained items at week 20. | Baseline, 20 weeks.
  Naming of ten trained phrases including an agent (subject), verb and a patient (object) with moving picture stimuli. Possible score ranges from 0 (worst) to 40 (best).

SECONDARY OUTCOMES:
Change from baseline in naming ability of untrained items at week 10. | Baseline, 10 weeks.
  A measure of generalization of treatment effects to naming of ten untrained phrases including an agent (subject), verb and a patient (object) with moving picture stimuli. Possible score ranges from 0 (worst) to 40 (best).
Change from baseline in naming ability of untrained items at week 20. | Baseline, 20 weeks.
  A measure of generalization of treatment effects to naming of ten untrained phrases including an agent (subject), verb and a patient (object) with moving picture stimuli. Possible score ranges from 0 (worst) to 40 (best).
Change from baseline in confrontation naming of single words (objects and actions) at week 10. | Baseline, 10 weeks.
  The Object & Action Naming Battery (Masterson & Druks, 1998) is a measure of change in ability to name forty pictures consisting of simple black and white drawings of objects and actions. Possible score range: 0 (worst) to 40 (best).
Change from baseline in confrontation naming of single words (objects and actions) at week 20. | Baseline, 20 weeks.
  The Object & Action Naming Battery (Masterson & Druks, 1998) is a measure of change in ability to name forty pictures consisting of simple black and white drawings of objects and actions. Possible score range: 0 (worst) to 40 (best).
Change from baseline in confrontation naming of single words (objects) at week 10. | Baseline, 10 weeks.
  The Boston naming test (Goodglass et al, 1983) is a measure of change in ability to name sixty simple black and white drawings of objects. Possible score range 0 (worst) to 60 (best).
Change from baseline in confrontation naming of single words (objects) week 20. | Baseline, 20 weeks.
  The Boston naming test (Goodglass et al, 1983) is a measure of change in ability to name sixty simple black and white drawings of objects. Possible score range 0 (worst) to 60 (best).
Change from baseline in connected speech at week 10. | Baseline, 10 weeks.
  Connected speech tasks (Nicholas & Brookshire, 1993) measures of change in ability to retrieve words in a picture description tasks, a procedural information task and in sharing personal information tasks. The speech produced in each task is analysed and number of words and adequate information units produced is calculated and related to time taken to produce the information. Higher numbers are better results.
Change from baseline in connected speech at week 20. | Baseline, 20 weeks.
  Connected speech tasks (Nicholas & Brookshire, 1993) measures of change in ability to retrieve words in a picture description tasks, a procedural information task and in sharing personal information tasks. The speech produced in each task is analysed and number of words and adequate information units produced is calculated and related to time taken to produce the information. Higher numbers are better results.
Change from baseline in self reported communicative participation in everyday life at week 10. | Baseline, 10 weeks.
  The Communicative Participation Item Bank (CPIB; Baylor et al 2013) is a validated measure of change in participants' perceptions of their communicative participation in everyday life activities. A short form of the item bank with ten items are used. The scoring of each item will be summarized into a total score with the range 0 (worse) to 30 (best).
Change from baseline in self reported communicative participation in everyday life at week 20. | Baseline, 20 weeks.
  The Communicative Participation Item Bank (CPIB; Baylor et al 2013) is a validated measure of change in participants' perceptions of their communicative participation in everyday life activities. A short form of the item bank with ten items are used. The scoring of each item will be summarized into a total score with the range 0 (worse) to 30 (best).
Change from baseline in self reported quality of life at week 10. | Baseline, 10 weeks.
  The Stroke Aphasia Quality of Life (SAQOL-39, Hilari et al 2009) is a validated measure of change in participant reported health related quality of life in a questionnaire with 39 items where participants evaluate of their everyday functioning in three domains: physical, psychosocial and communication. Scoring in each domain will be summarized and averaged and presented separately as well as in a compound averaged score. Possible score range is 1 (worse) to 5 (best).
Change from baseline in self reported quality of life at week 20. | Baseline, 20 weeks.
  The Stroke Aphasia Quality of Life (SAQOL-39, Hilari et al 2009) is a validated measure of change in participant reported health related quality of life in a questionnaire with 39 items where participants evaluate of their everyday functioning in three domains: physical, psychosocial and communication. Scoring in each domain will be summarized and averaged and presented separately as well as in a compound averaged score. Possible score range is 1 (worse) to 5 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Charlotta Saldert, Prof, Principal Investigator — Inst of Neurosci & Physiology, Speech & Language Pathology Unit, University of Gothenburg
Locations (1):
- University of Gothenburg, Västra Götalandsregionen, Gothenburg, Västra Götaland County, Sweden

REFERENCES:
- [Background] Baylor C, Yorkston K, Eadie T, Kim J, Chung H, Amtmann D. The Communicative Participation Item Bank (CPIB): item bank calibration and development of a disorder-generic short form. J Speech Lang Hear Res. 2013 Aug;56(4):1190-208. doi: 10.1044/1092-4388(2012/12-0140). Epub 2013 Jul 1. PMID 23816661
- [Background] Edmonds LA. Tutorial for Verb Network Strengthening Treatment (VNeST): Detailed Description of the Treatment Protocol with Corresponding Theoretical Rationale. Perspectives on Neurophysiology & Neurogenic Speech & Language Disorders. 2014; 24(3): 78-88
- [Background] Goodglass H, Kaplan E, Weintraub S. Boston Naming Test. Philadelphia, PA: Lea & Febiger. 1983.
- [Background] Hilari K, Lamping DL, Smith SC, Northcott S, Lamb A, Marshall J. Psychometric properties of the Stroke and Aphasia Quality of Life Scale (SAQOL-39) in a generic stroke population. Clin Rehabil. 2009 Jun;23(6):544-57. doi: 10.1177/0269215508101729. Epub 2009 May 15. PMID 19447841
- [Background] Long A, Hesketh A, Paszek G, Booth M, Bowen A. Development of a reliable self-report outcome measure for pragmatic trials of communication therapy following stroke: the Communication Outcome after Stroke (COAST) scale. Clin Rehabil. 2008 Dec;22(12):1083-94. doi: 10.1177/0269215508090091. PMID 19052247
- [Background] Masterson J, Druks J. Description of a set of 164 nouns and 102 verbs matched for printed word frequency, familiarity and age-of-acquisition. Journal of Neurolinguistics. 1998; 11: 331-54.
- [Background] Nicholas LE, Brookshire RH. A system for quantifying the informativeness and efficiency of the connected speech of adults with aphasia. J Speech Hear Res. 1993 Apr;36(2):338-50. doi: 10.1044/jshr.3602.338. PMID 8487525